CLINICAL TRIAL: NCT02610829
Title: Evaluation of a Short Course of Gamma Tocopherol Supplementation in Adult Subjects
Acronym: Gammadose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 15-1291; 5R01ES023349-03 (NIH)
Record Dates: First submitted 2015-11-06; First posted 2015-11-20 (Estimated); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: Gamma Tocopherol Serum Levels
MeSH Terms: interventions — gamma-Tocopherol; Vitamin E

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gamma Tocopherol (Experimental): Subjects will ingest 1400 mg gamma tocopherol, orally administered in 3 doses separated by 12 hours.
  Interventions: Dietary Supplement: Gamma tocopherol

INTERVENTIONS:
Dietary Supplement: Gamma tocopherol — 3 doses of 1400 mg gamma tocopherol (2 capsules, each is 700mg), at 12 hour intervals
  Other Names: Vitamin E

SUMMARY:
To evaluate serum levels of gamma tocopherol and it's metabolites after 3 doses, each separated by 12 hours.

DETAILED DESCRIPTION:
In previous studies the investigators have demonstrated that gamma-tocopherol-enriched (yT) supplementation decreased systemic oxidative stress, increased serum levels of yT, and inhibited monocyte responses to LPS without any adverse health effects. Free Radic Biol Med. 2008 Jul 1;45(1):40-9. doi: 10.1016/j.freeradbiomed.2008.03.002. Epub 2008 Mar 12.

Oxidant stress plays an important role in mucosal inflammation. Oxidant stress occurs individuals after exposure to air pollution, including high levels of ozone, LPS exposure and woodsmoke particle exposure. Potential exposure to all of these are naturally occurring events. Previous studies have also shown that asthmatic individuals tend to have lower endogenous levels of antioxidants such a s vitamins E and C, and that supplementing antioxidants can decrease exacerbation's associated with ozone exposure in children. The investigators are interested in future studies to examine the benefits of a rapid gamma tocopherol supplement in individuals who will be exposed to air pollution, either in a controlled chamber study or in a real life event, such as during high O3 days or when a woodsmoke fire is in their neighborhood.

This study is to address the question: can the investigators see an increase in serum levels of gT with a shorter course of gT supplementation? Additionally, before embarking on other investigations of gT as a potential prophylactic supplement, it is prudent to determine is discernible levels can be achieved with a shorter dose of gT.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between 18 and 50 years of age.
2. Vital signs within normal limits on admission to the study: SpO2 > 94%, systolic blood pressure between 150-90 mm Hg, diastolic blood pressure between 100-60 mm Hg, afebrile.

Exclusion Criteria:

1. Any chronic medical condition considered by the PI as a contraindication to receiving yT, including significant cardiovascular disease, diabetes requiring medication, chronic renal disease, chronic thyroid disease, kidney disease or coagulation defects.
2. Use of systemic or inhaled steroids.
3. Use of NSAID or ASA within 48 hours of dosing, and inability to withhold these medications for the duration of the study.
4. Use of anticoagulants including warfarin, heparin, clopidogrel or enoxaparin.
5. Diagnosis of anemia or abnormal blood counts at screening
6. Known vagal response to venipuncture
7. Abnormal PT or PTT values at screening.
8. BMI > 35
9. Pregnant or breast feeding women will not be included.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change in gamma tocopherol serum levels | Baseline, 30 hours after initial dosing

SECONDARY OUTCOMES:
Change in gamma-CEHC | Baseline, 30 hours after dosing initial dosing
Change in 5-NO-gamma tocopherol | Baseline, 30 hours after dosing initial dosing
Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment | Baseline, 30 hours after initial dosing

CONTACTS AND LOCATIONS:
Overall Officials: David B. Peden, MD, MS, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Center for Environmental Medicine, Asthma and Lung Biology, Chapel Hill, North Carolina, United States

REFERENCES:
- [Result] Wiser J, Alexis NE, Jiang Q, Wu W, Robinette C, Roubey R, Peden DB. In vivo gamma-tocopherol supplementation decreases systemic oxidative stress and cytokine responses of human monocytes in normal and asthmatic subjects. Free Radic Biol Med. 2008 Jul 1;45(1):40-9. doi: 10.1016/j.freeradbiomed.2008.03.002. Epub 2008 Mar 12. PMID 18405673